CLINICAL TRIAL: NCT03182868
Title: Vestibular Testing: Consistency and Effects Over Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Michael E. Hoffer, Professor of Otolaryngology, University of Miami
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 20150663
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Dizziness
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Repeatability Group (Experimental): Healthy participants perform goggle testing on two consecutive days to determine if the testing results are repeatable. Testing will be between 10 am and 2 pm and testing on the two sessions will be within 30 minutes of the same time. Sessions can be on two consecutive days or separated by up to 4 days.
  Interventions: Device: PAS Goggle
- Time of Day Group (Experimental): Healthy participants perform goggle testing at two different times of day to determine if time of day affects goggle testing performance. One quarter of the participants in this arm will undergo one test at 8 am on the first session and 10 am on the second session. A second quarter will undergo the tests at 10 am on first session and 8 am on the second session. A third quarter will undergo one test at 3 pm on the first session and 10 am on the second session. The fourth quarter will undergo the tests at 10 am on first session and 3 pm on the second session. In all these cases the sessions can be on consecutive days or separated by up to 4 days.
  Interventions: Device: PAS Goggle
- Learning Affect Group (Experimental): Healthy participants perform goggle testing back to back on the same day to determine if performance on second test changes from first test suggesting a learning affect.
  Interventions: Device: PAS Goggle
- MSQ Group (Experimental): Healthy participants perform goggle testing and upon completion of each goggle testing session will complete a Motion Sickness Questionnaire (MSQ) to determine if they show any signs of motion sickness.
  Interventions: Device: PAS Goggle
- OKN Only Group (Experimental): OKN Only Group is for exploratory aims only. Healthy participants will undergo goggle testing limited to Optokinetic Nystagmus (OKN) recordings at two stimulus speeds (20 and 60 deg/s) in both the counterclockwise and clockwise directions.
  Interventions: Device: PAS Goggle

INTERVENTIONS:
Device: PAS Goggle — PAS goggle is a self-contained stimulus and sensing device that is designed to deliver the visual stimuli currently delivered via light projected on a wall while simultaneously recording the movement of the eyes. Each vestibular testing session last about 15 minutes.

SUMMARY:
The goal of this study is to test the consistency and repeatability of a portable goggle system for testing optokinetic, ocular, and reaction time. The study examines the day to day consistency, time of day and learning effects as well as any secondary motion sickness.

DETAILED DESCRIPTION:
The goal of this study was to test the constancy and repeatability of this test by testing it in different individuals and different times of day, after a variety of tasks and after repeated performance

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* Both Females and males
* Staff and students at all levels at the University of Miami or first-degree - relatives/significant others of those individuals.

Exclusion Criteria:

* History of vestibular disorder/dysfunction
* Central processing disorder
* Impaired vision without corrective lenses (max 20/60 uncorrected)
* Moderate to severe hearing loss [>55 decibel (dB) Pure Tone Average (PTA), <50% word identification]

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-10-29 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoffer, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Repeatability Group | Time of Day Group | Learning Affect Group | MSQ Group | OKN Only Group
Started | 12 | 20 | 21 | 1 | 24
Completed | 9 | 20 | 17 | 0 | 16
Not Completed | 3 | 0 | 4 | 1 | 8
Not completed — Protocol Violation | 3 | 0 | 4 | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Repeatability Group | Time of Day Group | Learning Affect Group | MSQ Group | OKN Only Group | Total
Number analyzed (Participants) | 12 | 20 | 21 | 1 | 24 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 20 | 21 | 1 | 24 | 78
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 11 | 1 | 4 | 35
  Male | 5 | 8 | 10 | 0 | 20 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 4 | 4
  Unknown or Not Reported | 11 | 20 | 21 | 1 | 19 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 0 | 0 | 1 | 3 | 5
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 20 | 21 | 0 | 20 | 72

OUTCOME MEASURES:

1. Primary Outcome: Vestibular Reaction Times
Description: Repeatability, variation and learning effect of vestibular testing of PAS goggles will be evaluated using the test results on both sessions for the following sub-tests: a) Visual Reactive Time (VRT), b) Saccades and Reaction Time (SRT) Saccade Latency, c) SRT Motor Latency, and d) Auditory Reaction Time (ART). ART, VRT and SRT subtests are all evaluated in msec.
Time Frame: 2 Days
Population: Participants in the Repeatability, Time of Day and Learning Affect Groups were the only intended participants to be assessed for this outcome.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Repeatability Group | Time of Day Group | Learning Affect Group
Number analyzed (Participants) | 9 | 20 | 17
msec
  ART Session 1 | 240.89 (61.81) | 202.96 (41.43) | 233.09 (65.70)
  ART Session 2 | 228.95 (59.15) | 202.27 (57.42) | 213.07 (53.63)
  VRT Session 1 | 237.14 (47.89) | 212.21 (26.38) | 224.74 (42.22)
  VRT Session 2 | 229.52 (53.53) | 218.34 (30.73) | 230.63 (48.68)
  SRT Motor Latency Session 1 | 0.53 (0.11) | 0.41 (0.11) | 0.44 (0.14)
  SRT Motor Latency Session 2 | 0.49 (0.11) | 0.38 (0.11) | 0.44 (0.13)
  SRT Saccade Latency Session 1 | 0.20 (0.04) | 0.18 (0.03) | 0.20 (0.06)
  SRT Saccade Latency Session 2 | 0.18 (0.03) | 0.19 (0.03) | 0.20 (0.05)

2. Primary Outcome: Vestibular Subjective Visual Vertical
Description: Repeatability, variation and learning effect of vestibular testing of PAS goggles will be evaluated using the test results on both sessions for the Subjective Visual Vertical sub-test assessed in degrees.
Time Frame: 2 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Repeatability Group | Time of Day Group | Learning Affect Group
Number analyzed (Participants) | 9 | 20 | 17
degrees
  Session 1 | 2.08 (1.61) | 2.04 (2.36) | 1.21 (2.02)
  Session 2 | 1.52 (1.81) | 1.52 (2.17) | 1.64 (1.87)

3. Primary Outcome: Vestibular Smooth Pursuit Horizontal
Description: Repeatability, variation and learning effect of vestibular testing of PAS goggles will be evaluated using the test results on both sessions for the Smooth Pursuit Horizontal (SPH) sub-tests in degree squared per second.
Time Frame: 2 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degree squared per second
Arm/Group | Repeatability Group | Time of Day Group | Learning Affect Group
Number analyzed (Participants) | 9 | 20 | 17
degree squared per second
  Session 1 | 10006 (815) | 10739 (849) | 10303 (905)
  Session 2 | 9986 (754) | 10450 (818) | 10219 (1009)

4. Primary Outcome: Vestibular Percentage of Saccade
Description: Repeatability, variation and learning effect of vestibular testing of PAS goggles will be evaluated using the test results on both sessions for the sub-tests Smooth Pursuit Horizontal (SPH) evaluated as percentage of saccades completed.
Time Frame: 2 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Repeatability Group | Time of Day Group | Learning Affect Group
Number analyzed (Participants) | 9 | 20 | 17
percentage
  SPH Session 1 | 12.83 (12.14) | 16.49 (9.80) | 21.23 (13.70)
  SPH Session 2 | 12.72 (5.79) | 14.38 (8.38) | 18.23 (9.43)

5. Primary Outcome: Vestibular Anti-Saccade
Description: Repeatability, variation and learning effect of vestibular testing of PAS goggles will be evaluated using the test results on both sessions for the Anti-saccade sub-test evaluted in Percent Error.
Time Frame: 2 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of error
Arm/Group | Repeatability Group | Time of Day Group | Learning Affect Group
Number analyzed (Participants) | 9 | 20 | 17
percentage of error
  Session 1 | 39.09 (28.74) | 23.75 (17.16) | 34.56 (24.42)
  Session 2 | 28.17 (26.33) | 21.88 (15.11) | 24.26 (17.38)

6. Primary Outcome: Vestibular Gain
Description: Repeatability, variation and learning effect of vestibular testing of PAS goggles will be evaluated using the test results on both sessions for the following sub-tests: a) OKN at 60 degrees/second, and b) Smooth Percent Horizontal Velocity. Subtests are all evaluated in gain (output/input in decimal form)
Time Frame: 2 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Repeatability Group | Time of Day Group | Learning Affect Group
Number analyzed (Participants) | 9 | 20 | 17
ratio
  OKN Session 1 | 0.74 (0.09) | 0.78 (0.09) | 0.79 (0.09)
  OKN Session 2 | 0.72 (0.11) | 0.97 (0.07) | 0.77 (0.10)
  SPH Session 1 | 0.98 (0.04) | 0.74 (0.13) | 0.96 (0.06)
  SPH Session 2 | 0.99 (0.04) | 0.98 (0.08) | 0.95 (0.09)

7. Primary Outcome: Vestibular Saccade Horizontal
Description: Repeatability, variation and learning effect of vestibular testing of PAS goggles will be evaluated using the test results on both sessions for the Saccade Horizontal sub-tests evaluated in seconds.
Time Frame: 2 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Repeatability Group | Time of Day Group | Learning Affect Group
Number analyzed (Participants) | 9 | 20 | 17
seconds
  Session 1 | 0.17 (0.03) | 0.18 (0.02) | 0.18 (0.02)
  Session 2 | 0.18 (0.03) | 0.18 (0.02) | 0.18 (0.03)

8. Primary Outcome: Vestibular Predictive Saccade
Description: Repeatability, variation and learning effect of vestibular testing of PAS goggles will be evaluated using the test results on both sessions for the subtest Predictive Saccade (PS) evaluated as percentage of prediction.
Time Frame: 2 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of prediction
Arm/Group | Repeatability Group | Time of Day Group | Learning Affect Group
Number analyzed (Participants) | 9 | 20 | 17
percentage of prediction
  PS Session 1 | 37.04 (18.21) | 36.52 (21.99) | 35.88 (18.94)
  PS Session 2 | 32.66 (21.34) | 27.50 (20.79) | 35.12 (24.51)

9. Primary Outcome: Motion Sickness as Measured by the MSAQ
Description: Motion sickness is measured by the subjects being given a motion sickness assessment questionnaire (MSAQ). The MSAQ is a validated measure of motion sickness and in this questionnaire the examiner asks subjects 16 questions. Subjects score each question as "not at all" (score of zero) or on a seventy scale of 1-9. The total score ranging from 0-144 with the score reported as a percentage. The higher percentage score indicates more motion symptoms experienced by the subjects.
Time Frame: Day 1
Population: Participants in the MSQ Groups were the only intended participants to be assessed for this outcome. No participants completed the study for this arm.
Arm/Group | MSQ Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 days
Arm/Group | Repeatability Group | Time of Day Group | Learning Affect Group | MSQ Group | OKN Only Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/20 | 0/21 | 0/1 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/20 | 0/21 | 0/1 | 0/24
Other Adverse Events (participants affected / at risk) | 0/12 | 0/20 | 0/21 | 0/1 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No